CLINICAL TRIAL: NCT01294072
Title: Phase I Clinical Trial Investigating the Ability of Plant Exosomes to Deliver Curcumin to Normal and Malignant Colon Tissue
Brief Title: Study Investigating the Ability of Plant Exosomes to Deliver Curcumin to Normal and Colon Cancer Tissue
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Gerald W. Dryden, Jr., Professor, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: BCC-GI-10 Curcumin
Record Dates: First submitted 2011-02-03; First posted 2011-02-11 (Estimated); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Colon Cancer
Keywords: curcumin; plant exosomes; malignant colon tissue
MeSH Terms: conditions — Colonic Neoplasms | interventions — Curcumin

STUDY DESIGN:
Intervention Model Description: curcumin alone in capsule form (Arm 1) curcumin combined with plant exosomes (Arm 2) will not take curcumin or plant exosomes (Arm 3)
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1: Curcumin alone (Experimental): Subjects take curcumin orally.
  Interventions: Dietary Supplement: curcumin
- Arm 2: Curcumin with plant exosomes (Experimental): Subjects take curcumin conjugated with plant exosomes.
  Interventions: Dietary Supplement: Curcumin conjugated with plant exosomes
- Arm 3: no treatment (Experimental): subjects will not take curcumin or plant exosomes
  Interventions: Other: No intervention

INTERVENTIONS:
Dietary Supplement: curcumin — tablets-3.6 gram (gm) taken daily for 7 days - 15 subjects
  Arms: Arm 1: Curcumin alone
Dietary Supplement: Curcumin conjugated with plant exosomes — tablets-taken daily for 7 days - 15 subjects
  Arms: Arm 2: Curcumin with plant exosomes
Other: No intervention — no treatment
  Arms: Arm 3: no treatment

SUMMARY:
This clinical trial will investigate the ability of plant exosomes to more effectively deliver curcumin to normal colon tissue and colon tumors. Curcumin is the yellow pigment of turmeric, a natural product with diverse biological activities. Exosomes are small endosome-derived vesicles (50-100 nanometers [nm] in size). Previous clinical trials conducted with oral curcumin have demonstrated only limited bioavailability even at very high doses of 8-12 grams per day. This trial plans to address this problem of curcumin delivery by using plant exosomes to deliver the drug to colon tumors and normal colon tissue.

DETAILED DESCRIPTION:
Curcumin is a constituent of the spice turmeric, which is one of the primary ingredients of curry powder. Curcumin has been shown to interfere with colon carcinogenesis in a variety of chemical and genetic rodent models. It has also been shown to have a strong inhibitory effect on the growth of colon cancer cell lines. There is considerable evidence that the effects of curcumin are mediated by changes in signal transduction. There is an extensive body of work showing effects on several signaling pathways, including the beta-catenin and NF-κB pathways. Although curcumin has been viewed as an ideal chemopreventative agent in colon cancer for many years, its application has been impeded by important issues with drug delivery and bioavailability in the reported clinical trials of this compound.

Work from the James Graham Brown Cancer Center published recently suggests that using exosomes as a delivery vehicle leads to overcoming all the major obstacles of using curcumin as an anti-inflammatory agent, including increased stability, solubility, and bioavailability of curcumin. The work was further extended to define the resource that can supply a large quantity of exosomes with a maximum binding capacity of curcumin. Emerging data indicate that exosomes derived from many fruits release exosome-like particles, strongly bind to many hydrophobic drugs including curcumin, and are taken up by the intestine cells as well as the immune cells in the intestine. These results suggest that these fruit-derived exosomes are potentially used as a delivery vehicle to treatment of intestinal diseases. Moreover, both fruit exosomes and curcumin should not generate any side-effects since they are consumed by humans daily.

In this clinical trial, the effect of exosomally delivered curcumin on the immune modulation, cellular metabolism, and phospholipid profile of normal and malignant colon cells in subjects who are undergoing surgery for newly diagnosed colon cancer will be characterized. In selected subjects, the effect of exosomally delivered curcumin on the production of cytokines, the changes of immune cells, and glucose metabolism by administration of 13C-glucose prior to surgical resection will also be characterized.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have definitive diagnosis of colon cancer.
* Surgical resection of the primary tumor must be an option for the newly diagnosed cancer.
* No history of diabetes
* Subjects must be informed of the investigational nature of this study and sign and give written informed consent in accordance with institutional and federal guidelines.
* Absence of life-limiting medical conditions
* Ability to understand and willingness to sign a written informed consent document.
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2 (Karnofsky > 60%; see Appendix A).
* Subjects must have adequate bone marrow function. ANC > 1000/microliters (microL) and Platelet count >100,000/microL
* Age >20 years

Exclusion Criteria:

* Known familial colon cancer syndrome
* Pregnancy
* Known Human Immunodeficiency Virus (HIV)
* Patients receiving immunosuppressive drugs
* Inflammatory bowel disease
* Active second malignancy in the last 5 years
* Patients receiving any other investigational agent(s)
* Patients who have received any prior chemotherapy or radiation therapy to the primary colon cancer
* Intolerance to grapes, grapefruit, or curcumin
* History of diabetes mellitus

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2011-01; Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Concentration of curcumin in normal and cancerous tissue | 7 days after start of curcumin ingestion
  Concentration of curcumin delivered with curcumin alone or curcumin conjugated with plant exosomes to normal and cancerous colon cells will be compared. This exploratory trial is designed to estimate the effect of a fixed concentration of curcumin when delivered by plant exosomes compared to oral tablets of curcumin alone.

SECONDARY OUTCOMES:
safety and tolerability of curcumin alone as determined by adverse events | 7 days after study enrollment
  Curcumin will be taken orally.
effects of curcumin on normal and cancerous colon cells by measuring the biomarkers using histochemical staining | 7 days after patient enrollment
the immune system response to curcumin, measured by serum cytokine levels | 7 days after patient enrollment in study
immune response in ex vivo cell cultures of colon cancer cells treated with curcumin and Exo-cur, to be evaluated by using histochemical staining | 7 days after patient enrollment in study
measurement of curcumin alone on metabolic characteristics of normal colon mucosa and colon tumors | 7 days after patient enrollment
safety and tolerability of curcumin with plant exosomes as determined by adverse events | 7 days after study enrollment
  Curcumin and plant exosomes will be taken orally.
measurement of curcumin mixed with plant exosomes on metabolic characteristics of normal colon mucosa and colon tumors | 7 days after patient enrollment on study

CONTACTS AND LOCATIONS:
Overall Officials: Gerald W Dryden Jr, MD, PhD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville Hospital, Louisville, Kentucky, United States

REFERENCES:
- [Derived] Wu K, Xing F, Wu SY, Watabe K. Extracellular vesicles as emerging targets in cancer: Recent development from bench to bedside. Biochim Biophys Acta Rev Cancer. 2017 Dec;1868(2):538-563. doi: 10.1016/j.bbcan.2017.10.001. Epub 2017 Oct 18. PMID 29054476